CLINICAL TRIAL: NCT04554017
Title: Knowledge on Preventive Measures of Hypertension: An Interventional Study Among Senior High School Students, Kenyase - Ghana
Brief Title: Knowledge on Preventive Measures of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garden City University College (Other)
Responsible Party: Principal Investigator, Isaac Nkrumah, Lecturer, Garden City University College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DOS/VOL.2/01/2020/01
Record Dates: First submitted 2020-09-04; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm - All participant (Single arm) (Experimental): Participants received education or health talks on dietary and physical activity behaviours linked to hypertension
  Interventions: Other: Education/Training

INTERVENTIONS:
Other: Education/Training — It consisted of a brief overview of hypertension, risk factors, complications and much emphasis placed on the preventive measures (what they include and why it is necessary to practice them).

SUMMARY:
Hypertension among children and adolescents is on the rise in both developed and developing countries. Childhood and adolescent obesity, a key factor for hypertension in this population results largely from unhealthy dietary and physical inactivity behaviours. Adequate knowledge, a component for behavior change, has been found to be crucial to improving one's confidence to tackle these improper behaviours. Despite this, there are gaps in knowledge on hypertension and its risks factors in Ghanaian adolescents. Using an educational intervention (health talk), the study therefore sought to improve knowledge on preventive measures of hypertension among senior high school students in Ghana.

DETAILED DESCRIPTION:
A pre-post interventional study using health talks was carried out among 345 adolescents aged 13 to 20 years. Participants included both male and female students aged 13 to 20 years. Owing to the large number, the students were divided into two groups. The Pre-test was then administered. Following this, two health education sessions were delivered by two registered nurses for each session. A week after these health talks, the research team went back to the school to collect data for the post-intervention. Questionnaires used for both pre and post assessment collected data on demographic factors and knowledge on dietary and physical activity behaviours linked to hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants who gave consent
* Minors with parental or guardian assent

Exclusion Criteria:

* Participants already living with hypertension

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 345 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Change in participants knowledge on the preventives measures of hypertension using the mean scores | 1 week
  Close ended questionnaire was used to assess participants' knowledge on dietary practices and physical activity related to prevention of hypertension. The same questions were administered both pre- and post-assessment

SECONDARY OUTCOMES:
Association between the demographic characteristics and impact of the educational intervention on adolescents' knowledge on the preventive measures was measured using logistic regression analysis | 1 week
  In order to determine the association between the demographic characteristics and the impact of education on student's knowledge, the mean change in knowledge was categorize into two: <50% impact and ≥50%. Significance was set at p-value < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Nkrumah, Masters, Principal Investigator — Garden City University College
Locations (1):
- Isaac Nkrumah, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made availability online immediately the paper is published in a journal. This will however, be before 12 months following study completion
Supporting Information: Study Protocol, ICF
Time Frame: immediately the paper is published - before 12 months following study completion
Access Criteria: online or using the web address by the published journal